CLINICAL TRIAL: NCT04953208
Title: The DiSCoVeR Project: Examining the Synergistic Effects of a Cognitive Control Videogame and a Self-administered Non-invasive Brain Stimulation on Alleviating Depression
Brief Title: Remotely Non-invasive Brain Stimulation and Videogame to Alleviate Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mor Nahum (Other)
Collaborators: Hadassah Medical Organization (Other); Ludwig-Maximilians - University of Munich (Other); Riga Stradins University (Other)
Responsible Party: Sponsor-Investigator, Mor Nahum, Principal Investigator, Hebrew University of Jerusalem
Organization: Hebrew University of Jerusalem (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 388-20-HMO
Record Dates: First submitted 2021-06-07; First posted 2021-07-07 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
Keywords: cognitive control; non-invasive brain stimulation, transcranial direct current stimulation; VideoGame; self-application; home-based; feasibility; efficacy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): active tDCS (using the Neuroelectrics Starstim tCS 5G kit) and cognitive and emotional control video game
  Interventions: Device: active tDCS; Behavioral: cognitive and emotional control video game
- Sham treatment (Sham Comparator): sham tDCS (using the Neuroelectrics Starstim tCS 5G kit) and non-active videogame
  Interventions: Device: sham tDCS; Behavioral: sham video game

INTERVENTIONS:
Device: active tDCS — Treatment will be applied daily 5 days/week for a period of 6 weeks, which equals a tDCS stimulation for a total of 30 treatment sessions. Every treatment session consists of 30 minutes of intervention.
  Arms: Active treatment
Device: sham tDCS — sham stimulation for a total of 30 treatment sessions. Every treatment session consists of 30 minutes of intervention.
  Arms: Sham treatment
Behavioral: cognitive and emotional control video game — a video game targeting cognitive and emotional control. total of 30 treatment sessions. Every treatment session consists of 30 minutes of intervention.
  Arms: Active treatment
Behavioral: sham video game — a video game which does not target cognitive control, played for total of 30 treatment sessions. Every treatment session consists of 30 minutes of intervention.
  Arms: Sham treatment

SUMMARY:
Major depressive disorder (MDD) is a common, recurrent, and frequent chronic disorder. Treatment is often challenging; up to 40% of patients do not benefit sufficiently from existing antidepressant interventions including trials of medication and psychotherapy. Up to 25% of patients manifest a chronic course of illness, resulting in a need for additional treatment options.

The DiSCoVeR trial is a multi-site, double-blind, sham-controlled, proof-of concept randomized controlled trial (RCT). The study aims to investigate the feasibility and efficacy of an innovative, combined treatment approach, incorporating transcranial direct current stimulation (tDCS) along with a custom-made video game designed to enhance cognitive control in patients with major depressive disorder (MDD).

Patients diagnosis of MDD receive a 6-weeks treatment with prefrontal tDCS along with an active videogame or sham tDCS + sham game for 6 weeks. Follow-up per patient is 6 weeks following treatment. Before, during and after the treatment period different assessment scales will be conducted to record neuropsychological features and the course of symptom changes.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a prevalent, seriously impairing, and often recurrent mental disorder. It has been ranked as a leading cause of disability worldwide by the World Health Organization (WHO) as measured by years lived with disability.

A considerable number of patients with MDD experience a chronic course of illness and approximately one third of MDD patients do not respond sufficiently to pharmacological treatment, calling for treatment alternatives.

Non-invasive brain stimulation techniques (NIBS) such as tDCS targeting prefrontal cortical areas have emerged as a safe, promising, and cost-effective alternative to traditional treatment options in patients with MDD.

This study focuses not only on an overall reduction of depressive symptoms, but also an alleviation of cognitive control deficits in particular, since patients with MDD often suffer from cognitive control deficits. tDCS has been shown to directly modulate cognitive control functions in healthy participants and in depressed patients. Another approach to directly modulate cognitive control functions is cognitive control training.

In the present study, an engaging and captivating cognitive control training designed as an action video game will be employed. The primary objective is to test the feasibility and efficacy of this innovative, combined treatment approach for self application, concurrently applying both interventions (tDCS + cognitive control training) in patients suffering from MDD. Additionally, participants have the opportunity to choose to take part in two adjunctive assessments: a biological assessment which includes salivary samples and a multimodal imaging paradigm (structural and functional sequences, including an interleaved TMS-fMRI paradigm).

ELIGIBILITY:
Inclusion criteria:

* Men and woman 18-65 years of age.
* Primary Diagnostic and Statistical Manual (DSM-5) diagnosis of Major Depressive Disorder (MDD), with a single or recurrent episode with the additional requirement of a current episode with a duration of ≥4 weeks.
* Current depressive episode lasts less than 5 years (the current and previous depressive episodes are demarcated by a period of ≥2 months in which the patient did not meet full criteria for the DSM-5 definition of MDD).
* Total Hamilton-21 score ≥ 13 at screening visit.
* Capable and willing to provide informed consent. Patients without antidepressant medication or patients on an adequate (i.e., at least lowest effective) and stable (i.e., for ≥ 6 weeks) dosage of SSRI (Escitalopram, Citalopram, Sertralin, Paroxetin, Fluvoxamin, Fluoxetin), SSNRI (Duloxetin, Venlafaxin) or Others (Mirtazapin, Agomelatin, Vortioxetine)
* Concomitant psychotherapy is allowed if ongoing for at least 3 months prior to baseline.

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption).
* Addiction to gaming as assessed by the Gaming Disorder Test (GDT).
* Individuals diagnosed with the following psychiatric conditions (current unless otherwise stated):

  * Depression assessed as secondary to a general medical condition or substance-induced
  * Substance abuse or substance dependence (except nicotine, caffeine) in the last 6 months
  * Psychotic disorder (lifetime)
  * Bipolar disorder (I and II; lifetime)
  * Eating disorder if stated as primary diagnosis
  * Obsessive compulsive disorder if stated as primary diagnosis
  * Post-traumatic stress disorder if stated as primary diagnosis
  * Generalized anxiety disorder if stated as primary diagnosis
  * Panic disorder/ social anxiety if stated as primary diagnosis
  * Personality disorder if stated as primary diagnosis
* Individuals diagnosed with a significant neurological disorder or insult including, but not limited to:

  * Increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm, dementia
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
  * Epilepsy
* Electroconvulsive therapy (ECT) treatment in current episode
* History of tDCS, except for single tDCS sessions in experimental studies
* Use of any investigational drug within 6 weeks from baseline
* Suicidal risk based on MADRS item 10 score of 4-6 or attempted suicide in current episode
* Acute, unstable cardiac disease
* Intracranial implant or any other metal object within or near the head (excluding the mouth) that cannot be safely removed; implanted neuro-stimulators
* Known or suspected pregnancy (according to pregnancy test), and women of childbearing potential not using effective contraception
* History of seizures
* Treatment with deep brain stimulation or vagus nerve stimulation and/or any other intracranial implants (clips, cochlear implants)
* Any relevant unstable medical condition (e.g. acute, unstable cardiac disease)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of treatment | Six weeks
  Feasibility is met if a patient will complete 20 sessions per protocol with a probability of more than 50.00%.Completion per protocol is achieved, if the patient completes 20 sessions per protocol with a probability of more than 50 percent.

SECONDARY OUTCOMES:
Efficacy-Improvement on the MADRS scores compared to baseline. | six weeks
  Change from baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) scores at week 6 post-randomization compared to baseline.
  The MADRS scores severity of depression on a scale from 0-60. Higher scores indicate worse depression. A total score between 0-6 indicates that the patient is in the normal range (no depression), 7-19 indicates mild depression, 20-34 indicates moderate depression, and a score of 35 and greater indicates severe depression.

CONTACTS AND LOCATIONS:
Locations (3):
- Ludwig-Maximilian University, Munich, Germany
- Hadassah University Hospital, Jerusalem, Israel
- Riga Stradins University (RSU), Riga, Latvia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Padberg F, Bulubas L, Mizutani-Tiebel Y, Burkhardt G, Kranz GS, Koutsouleris N, Kambeitz J, Hasan A, Takahashi S, Keeser D, Goerigk S, Brunoni AR. The intervention, the patient and the illness - Personalizing non-invasive brain stimulation in psychiatry. Exp Neurol. 2021 Jul;341:113713. doi: 10.1016/j.expneurol.2021.113713. Epub 2021 Mar 31. PMID 33798562
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Stewart JW, Nierenberg AA, Thase ME, Ritz L, Biggs MM, Warden D, Luther JF, Shores-Wilson K, Niederehe G, Fava M; STAR*D Study Team. Bupropion-SR, sertraline, or venlafaxine-XR after failure of SSRIs for depression. N Engl J Med. 2006 Mar 23;354(12):1231-42. doi: 10.1056/NEJMoa052963. PMID 16554525
- [Result] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871
- [Result] Padberg F, Kumpf U, Mansmann U, Palm U, Plewnia C, Langguth B, Zwanzger P, Fallgatter A, Nolden J, Burger M, Keeser D, Rupprecht R, Falkai P, Hasan A, Egert S, Bajbouj M. Prefrontal transcranial direct current stimulation (tDCS) as treatment for major depression: study design and methodology of a multicenter triple blind randomized placebo controlled trial (DepressionDC). Eur Arch Psychiatry Clin Neurosci. 2017 Dec;267(8):751-766. doi: 10.1007/s00406-017-0769-y. Epub 2017 Feb 28. PMID 28246891
- [Result] De Raedt R, Koster EH. Understanding vulnerability for depression from a cognitive neuroscience perspective: A reappraisal of attentional factors and a new conceptual framework. Cogn Affect Behav Neurosci. 2010 Mar;10(1):50-70. doi: 10.3758/CABN.10.1.50. PMID 20233955
- [Result] Wolkenstein L, Plewnia C. Amelioration of cognitive control in depression by transcranial direct current stimulation. Biol Psychiatry. 2013 Apr 1;73(7):646-51. doi: 10.1016/j.biopsych.2012.10.010. Epub 2012 Dec 6. PMID 23219367
- [Result] Calkins AW, McMorran KE, Siegle GJ, Otto MW. The Effects of Computerized Cognitive Control Training on Community Adults with Depressed Mood. Behav Cogn Psychother. 2015 Sep;43(5):578-89. doi: 10.1017/S1352465814000046. Epub 2014 Mar 3. PMID 24589123
- [Result] Bavelier D, Green CS. Enhancing Attentional Control: Lessons from Action Video Games. Neuron. 2019 Oct 9;104(1):147-163. doi: 10.1016/j.neuron.2019.09.031. PMID 31600511
- [Result] Hoorelbeke K, Koster EHW. Internet-delivered cognitive control training as a preventive intervention for remitted depressed patients: Evidence from a double-blind randomized controlled trial study. J Consult Clin Psychol. 2017 Feb;85(2):135-146. doi: 10.1037/ccp0000128. Epub 2016 Jun 30. PMID 27362792
- [Derived] Dechantsreiter E, Padberg F, Morash A, Kumpf U, Nguyen A, Menestrina Z, Windel F, Burkhardt G, Goerigk S, Morishita T, Soldini A, Ahissar S, Cohen T, Pasqualotto A, Rubene L, Konosonoka L, Keeser D, Zill P, Assi R, Gardier R, Vinals R, Thiran JP, Segman R, Benjamini Y, Bonne O, Hummel FC, Bavelier D, Rancans E, Nahum M. Examining the synergistic effects of a cognitive control video game and a home-based, self-administered non-invasive brain stimulation on alleviating depression: the DiSCoVeR trial protocol. Eur Arch Psychiatry Clin Neurosci. 2023 Feb;273(1):85-98. doi: 10.1007/s00406-022-01464-y. Epub 2022 Oct 22. PMID 36271928